CLINICAL TRIAL: NCT04291469
Title: A Prospective, Randomized, Controlled Multicenter Trial of Probiotics and Prebiotics to Improve the Efficacy of Antipsychotics in Patients With Schizophrenia
Brief Title: Antipsychotic Effects of Probiotics and Prebiotics on Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: BaoJi Rehabilitation Hospital (Unknown); Xiangyang Central Hospital (Other); WeiNan Psychiatry Hospital (Unknown); HanZhong Psychiatric Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2019-003
Record Dates: First submitted 2020-02-13; First posted 2020-03-02 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Probiotics
MeSH Terms: conditions — Schizophrenia | interventions — Lacteol; Prebiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Identical-appearing Placebo (maltodextrin tables) ,oral, daily for 14 weeks
  Interventions: Dietary Supplement: maltodextrin
- Probiotics group (Experimental): Combined Bifidobacteria+lactobacillus+maltodextrin tables, each table contain more than 1.0*10^9 colony forming units, oral, daily for 14 weeks
  Interventions: Drug: Probiotics（Live combined bifidobacteria, lactobacillus and maltodextrin tables)
- Prebiotics group (Experimental): Combined inulin+maltodextrin tables, oral, daily for 14 weeks
  Interventions: Dietary Supplement: Prebiotics (Combined inulin and maltodextrin tables)

INTERVENTIONS:
Drug: Probiotics（Live combined bifidobacteria, lactobacillus and maltodextrin tables) — The probiotic compound will consist of tables containing approximately 10^9 colony forming units of the probiotic organisms, Lactobacillus and Bifidobacteria lactis strain，mixed maltodextrin(oral, daily for 14 weeks).
  Other Names: Probiotic bacteria
  Arms: Probiotics group
Dietary Supplement: Prebiotics (Combined inulin and maltodextrin tables) — The prebiotic compound will consist of tables containing inulin and maltodextrin (oral,daily for 14 weeks)
  Arms: Prebiotics group
Dietary Supplement: maltodextrin — Maltodextrin tables (oral,daily for 14 weeks)
  Arms: Control group

SUMMARY:
In this study, investigators will evaluate the efficacy and related mechanism of probiotics and prebiotics as an add-on treatment in improving the antipsychotic induced psychotic syndrome, the cognitive impairment, gastrointestinal function, and metabolic disorders in schizophrenia patients, through genotype identification, psychopathology, neuropsychology, biochemical evaluation and other methods.

DETAILED DESCRIPTION:
The study will recruit 210 schizophrenia patients who meet the criteria of DSM-4, and then randomized to 3 groups: control group, probiotics group and prebiotics group for a 14-weeks clinical trail and 12-weeks follow-up period. In addition to probiotics, prebiotic or maltodextrin interventions, in the meantime, all participants will also use one of the prescribed antipsychotics medications. Clinical efficacy and safety assessment will be done at baseline, clinical trail and follow-up period. The specific aims are to evaluate these tips: 1) psychotic syndrome; 2) cognition; 3) Gastrointestinal function; 4) inflammatory and metabolic related markers. Psychotic syndrome will be measured by the Positive and Negative Syndrome Scale. Cognitive function will be assessed by the MATRICS Consensus Cognitive Battery. Gastrointestinal function will be assessed by gastrointestinal symptom assessment scale (GSRS). Biological samples also will be collected, and stored to research Intestinal inflammation, intestinal permeability, intestinal flora and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Diagnostic and Statistical Manual (DSM-V) diagnostic criteria for schizophrenia
* Duration of illness 5 years, Subjects are currently receiving first-line recommended antipsychotic medication
* The total PANSS score ≥60, containing at least three positive or negative items with scores of 3 or more at screening
* Junior high school or above
* Capacity for written informed consent.

Exclusion Criteria:

* Pregnant or lactating women
* Any clinically significant or unstable medical disorder as determined by the investigators, including congestive heart failure, abnormal liver function, renal failure, immunodeficiency diseases, cancer, or gastrointestinal diseases ( inflammatory bowel disease or celiac disease, except functional constipation)
* Subjects had acute or chronic infections or are taking anti-inflammatory drugs and cortisol hormones. Receipt of antibiotic medication within the previous 1 month.
* Other neuropsychiatric disorders (organic diseases of the central nervous system, a mental disorder caused by a physical disease or psychoactive substance, mental retardation).
* Having history of substance dependence or abuse，including alcohol
* BMI is not within the normal range (18.5 to 23.9)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) Score from week0 to week26 | 26weeks(week0 to week26)
  The complete PANSS contains ratings for 30 symptoms, including 7 positive symptoms, 7 negative symptoms, and 16 general psychiatric symptoms. The clinical efficacy was evaluated by its score reduction rate, with the total score reduction rate ≥75% as recovery, 50% ~ 74% as significant improvement, 25% ~ 49% as improvement, and <25% as invalid. improvement, significant improvement and recovery add up to apparent effect.

SECONDARY OUTCOMES:
Change in MATRICS Consensus Cognitive Battery(MCCB) Score from week1 to week26 | week26(week1 to week26 )
  Change in the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) score from the start of Trial period to the end of the follow-up phase; Cognitive performance is measured by the MATRICS Consensus Cognitive Battery composite score in participants.
Gastrointestinal symptom rating scale (GSRS) | week26 (week1 to week26)
  Gastrointestinal function will be assessed during the screening stage，week 4, week 8, week 12, week 14 of treatment stage and once every 4 weeks of follow-up stage through Gastrointestinal symptom rating scale (GSRS); The score reduction of GSRS≥25% was associated with improvement in gastrointestinal function.
Serum inflammatory factors-TH-1 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --TH-1
Serum inflammatory factors-TH-2 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines--TH-2
Serum inflammatory factors-TH-17 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines--TH-17
Serum inflammatory factors-Interleukin-1 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines--Interleukin-1
Serum inflammatory factors-Interleukin-2 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --Interleukin-2
Serum inflammatory factors-Interleukin-6 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --Interleukin-6
Serum inflammatory factors-Interleukin-10 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --Interleukin-10
Serum inflammatory factors-Interleukin-17 | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --Interleukin-17
Serum inflammatory factors-TNF-a | week26(week1 to week26)
  Change of intestinal inflammation will be assessed during the the double-blind phase, including serum inflammatory cytokines --TNF-a(tumor necrosis factor-a,interferon).
Fecal intestinal flora | week26 (week1 to week26)
  The number of lactobacillus and bifidobacterium flora will be assessed; The species and abundance of intestinal flora were identified by 16SrRNA.
Serum intestinal permeability index-FABP2 | week26(week1 to week26)
  Change of Serum intestinal permeability index will be assessed during the the double-blind phase- FABP2
Serum intestinal permeability index-sCD14 | week26(week1 to week26)
  Change of Serum intestinal permeability index will be assessed during the the double-blind phase-sCD14
Serum intestinal permeability index-LBP | week26(week1 to week26)
  Change of Serum intestinal permeability index will be assessed during the the double-blind phase-LBP

CONTACTS AND LOCATIONS:
Overall Officials: Xiancang Ma, M.D., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiao tong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
If necessary, part of the data can be obtained through the project leader.